CLINICAL TRIAL: NCT07254832
Title: No Significant Alterations in Balance Performance After Acute Caffeine and Nicotine Gum Intake in Trained Athletes
Brief Title: Effects of Caffeine and Nicotine Gum on Balance Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gülbin Rudarlı (Other)
Responsible Party: Sponsor-Investigator, Gülbin Rudarlı, Professor of Sport Sciences, Department of Coaching Education, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EGE-24-3.1T-81
Record Dates: First submitted 2025-07-08; First posted 2025-11-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Athletic Performance; Postural Stability; Healhty
Keywords: Caffeinated chewing gum; Nicotine chewing gum; Caffeine; Nicotine; Dynamic balance; Postural control; Ellipse area; Perimeter length; Trained athletes
MeSH Terms: interventions — Nicotine Chewing Gum; Xylitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- caffeine gum (Experimental)
  Interventions: Dietary Supplement: Caffeine Gum 3mg/kg
- Nicotine Gum (Active Comparator)
  Interventions: Dietary Supplement: Nicotine Gum (4 mg)
- Placebo Gum (Placebo Comparator)
  Interventions: Other: Placebo Gum (Xylitol)
- Control (No Intervention): No chewing gum administered; participants completed balance testing without any intervention.

INTERVENTIONS:
Dietary Supplement: Caffeine Gum 3mg/kg — Participants chewed 2-3 pieces of 100 mg caffeine gum (~3 mg/kg total) for 5 minutes prior to balance testing.
  Arms: caffeine gum
Dietary Supplement: Nicotine Gum (4 mg) — Participants chewed one piece of 4 mg nicotine gum for 30 minutes before undergoing balance testing.
  Arms: Nicotine Gum
Other: Placebo Gum (Xylitol) — Participants chewed xylitol-based sugar-free gum with no active substance for 20 minutes prior to testing.
  Arms: Placebo Gum

SUMMARY:
This randomized, single-blind, placebo-controlled, four-condition crossover study evaluates the acute effects of caffeine gum (~3 mg/kg) and nicotine gum (4 mg) on balance performance in healthy, trained adults. Each participant completes four test visits (caffeine gum, nicotine gum, xylitol-based placebo gum, and no-gum control) separated by ≥24 hours. Static and dynamic balance are assessed using the ProKin 252 system under standardized procedures. The primary outcomes are postural sway (ellipse area) and center-of-pressure path length over predefined test trials/time frames. The objective is to determine whether acute administration of these stimulants alters balance-related performance relative to placebo and control.

DETAILED DESCRIPTION:
This study evaluates the acute effects of two commonly used stimulants-caffeine and nicotine administered in chewing-gum form-on static and dynamic balance performance in healthy, trained adults. The trial uses a randomized, single-blind, placebo-controlled, four-condition crossover design. Twenty participants complete four laboratory visits scheduled at the same time of day and separated by a washout interval of at least 24 hours. The order of the four conditions is randomized.

Interventions are: (1) caffeine gum at approximately 3 mg/kg, (2) nicotine gum at 4 mg, (3) sugar-free xylitol-based placebo gum, and (4) a no-gum control condition. Pre-testing exposure is standardized across conditions: caffeine gum is chewed for 5 minutes, nicotine gum for 30 minutes, and placebo gum for 20 minutes prior to balance assessments. The control condition involves no gum exposure. All procedures are conducted under uniform laboratory conditions.

Balance performance is assessed immediately after the pre-specified exposure period using the ProKin 252 balance platform. Standardized static and dynamic balance tasks are administered according to device guidelines and site procedures. Primary outcomes are postural sway quantified as ellipse area and center-of-pressure path length over predefined trials/time frames. Additional procedural details (e.g., task sequence, rest intervals, and device settings) are maintained in the study manual to ensure consistency across visits.

The objective is to determine whether acute administration of caffeine or nicotine, relative to placebo and control, alters balance-related performance indices in healthy, physically active individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Be healthy, with no diagnosed neurological or musculoskeletal disorders
2. Be physically active and have at least 3 years of regular training history
3. Be between 18 and 30 years of age
4. Have no balance impairments or vestibular issues
5. Be non-smoker or not using tobacco during study days
6. Able to comply with the intervention protocols and attend all test sessions
7. Provide written informed consent

Exclusion Criteria:

1. Training age less than three years,
2. Having a disease or sports injury that will affect balance performance,
3. Using a drug or substance that affects balance,
4. Not being able to comply with or continue the study measurements.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Static Postural Sway Ellipse Area - ProKin 252 Stabilometric Platform | At each visit: 5 minutes after start of chewing (caffeine gum), 30 minutes after start of chewing (nicotine gum), 20 minutes after start of chewing (xylitol placebo gum), and 0 minutes (no gum) for the control condition; single 30-second trial per visit
  Center of pressure (COP) 95% ellipse area during quiet bipedal stance (eyes open; standardized foot position) measured with the ProKin 252. Higher values indicate poorer balance.
  Unit of Measure: mm^2

SECONDARY OUTCOMES:
Static Center of Pressure (COP) Path Length - ProKin 252 Stabilometric Platform | At each visit: 5 minutes after start of chewing (caffeine gum), 30 minutes after start of chewing (nicotine gum), 20 minutes after start of chewing (xylitol placebo gum), and 0 minutes (no gum) for the control condition; single 30-second trial per visit
  Total COP excursion length during quiet bipedal stance (eyes open; standardized foot position) measured with the ProKin 252. Higher values indicate poorer balance.
  Unit of Measure: mm

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Faculty of Sport Sciences, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No